CLINICAL TRIAL: NCT02019225
Title: Time to Reduce Mortality in End-Stage Renal Disease (TiME) Trial
Brief Title: A Cluster-randomized, Pragmatic Trial of Hemodialysis Session Duration
Acronym: TiME
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient separation in session duration between randomized treatment groups
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institutes of Health (NIH) (NIH); Fresenius Medical Care North America (Industry); Davita Clinical Research (Industry); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 817911; UH3DK102384 (NIH); UH2AT007797 (NIH)
Record Dates: First submitted 2013-10-30; First posted 2013-12-24 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: End Stage Renal Disease
Keywords: dialysis; hemodialysis; pragmatic trial; end stage renal disease; randomized clinical trial
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dialysis session of at least 4.25 hours (Experimental): Dialysis facilities randomized to the Intervention arm will adopt an approach of recommending that all patients who are initiating treatment with maintenance hemodialysis have a treatment session duration of at least 4.25 hours.
  Interventions: Other: Dialysis session of at least 4.25 hours
- Usual care (No Intervention): There will be no trial-driven approach to dialysis session duration in the Usual Care arm.

INTERVENTIONS:
Other: Dialysis session of at least 4.25 hours — Facilities randomized to the Intervention arm will adopt the practice of recommending dialysis session durations of at least 4.25 hours for all patients initiating hemodialysis treatment regardless of body size or dialysis solute clearance measurements.
  Arms: Dialysis session of at least 4.25 hours

SUMMARY:
The purpose of the TiME Trial is to determine whether dialysis facility implementation of a minimum hemodialysis session duration of 4.25 hours (versus usual care) for patients with end-stage renal disease initiating treatment with thrice weekly maintenance hemodialysis has benefits on mortality, hospitalizations and health-related quality of life.

The trial also aims to demonstrate the capacity to conduct a large, pragmatic clinical trial in partnership with two large dialysis provider organizations.

DETAILED DESCRIPTION:
The TiME Trial is a cluster-randomized, parallel-group pragmatic clinical trial for patients initiating treatment with maintenance hemodialysis. Facilities will be randomized in a 1:1 distribution to the Intervention arm or the Usual Care arm. Facilities randomized to the Intervention arm will adopt the practice of recommending dialysis session durations of at least 4.25 hours for all patients initiating hemodialysis treatment regardless of body size or dialysis solute clearance measurements. Facilities randomized to Usual Care will maintain their existing approaches to prescribing dialysis session duration. Participants will be followed for up to 3 years. The primary endpoint is mortality; major secondary endpoints are hospitalization rate and quality of life. Pragmatic features of the TiME Trial include 1) high generalizability due to non-restrictive eligibility criteria and broad representation of participating facilities, 2) implementation of the intervention by clinical care providers rather than by research personnel, and 3) reliance on data obtained through routine clinical care rather than through research activities.

ELIGIBILITY:
Inclusion Criteria: End stage renal disease patients treated by hemodialysis on a thrice weekly maintenance schedule:

* Initiation of maintenance dialysis within the past 120 days.
* Treatment with maintenance dialysis in a participating facility.
* Age ≥18 years.

Exclusion Criteria:

* Unwillingness to participate.
* Inability to provide consent for dialysis care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7053 (Actual)
Dates: Start 2013-12-18 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
All cause mortality | Throughout the 3 year (maximum) duration of follow-up
  The primary outcome for the TiME Trial is time to death. The trial hypothesis is that, in comparison with the Usual Care facilities, the risk of death will be lower in the facilities randomized to the Intervention group.

SECONDARY OUTCOMES:
Hospitalization rate | Throughout the 3 year (maximum) duration of follow-up
  Hospitalization rate is a major secondary outcome of the TiME Trial. The trial hypothesis is that, in comparison with the Usual Care facilities, the rate of hospitalization will be lower in the facilities randomized to the Intervention group.

OTHER OUTCOMES:
Quality of Life | Annually throughout the duration of follow-up. Patients will be followed up to 3 years.
  The Health Related Quality of Life (HRQOL) questionnaire used for the TiME Trial will be the KDQOL™36, a kidney disease-specific instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Dember, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Fresenius Medical Care North America, Waltham, Massachusetts
  - DaVita Clinical Research, Minneapolis, Minnesota

REFERENCES:
- [Derived] Johnson KE, Neta G, Dember LM, Coronado GD, Suls J, Chambers DA, Rundell S, Smith DH, Liu B, Taplin S, Stoney CM, Farrell MM, Glasgow RE. Use of PRECIS ratings in the National Institutes of Health (NIH) Health Care Systems Research Collaboratory. Trials. 2016 Jan 16;17:32. doi: 10.1186/s13063-016-1158-y. PMID 26772801